CLINICAL TRIAL: NCT02664961
Title: A Phase 2A Study of TRC105 (With Option to Add Bevacizumab) in Patients With Refractory Gestational Trophoblastic Neoplasia (GTN)
Brief Title: Study of TRC105 and Bevacizumab in Patients With Refractory Gestational Trophoblastic Neoplasia (GTN)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Rare tumor type, patients eligible via expanded access.
Sponsor: Tracon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105GTN201
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-05

CONDITIONS: Gestational Trophoblastic Neoplasia; Choriocarcinoma; Placental Site Trophoblastic Tumor; Epithelioid Trophoblastic Tumor
Keywords: TRC105; CD105; Endoglin; Angiogenesis inhibitor; GTN; Bevacizumab; Avastin
MeSH Terms: conditions — Gestational Trophoblastic Disease; Choriocarcinoma; Trophoblastic Tumor, Placental Site | interventions — carotuximab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRC105 and/or bevacizumab (Experimental): All subjects will begin by receiving single agent TRC105 weekly. In the case of a complete response to single agent TRC105, subjects will continue to receive single agent TRC105 for at least 3 months following complete response. In the case of a partial response (without a complete response) to single agent TRC105, bevacizumab every two weeks will be added. In the absence of a partial or complete response to single agent TRC105, subjects will receive single agent bevacizumab every two weeks. In the absence of a complete response to single agent bevacizumab, or for subjects who have documented disease progression on a prior bevacizumab containing regimen, subjects will receive TRC105 weekly and bevacizumab every two weeks.
  Interventions: Drug: TRC105; Drug: Bevacizumab

INTERVENTIONS:
Drug: TRC105 — Subjects will begin by receiving TRC105 weekly. Subjects who achieve a complete response on single agent TRC105 may transition to every two week dosing.
  Other Names: Chimeric Antibody (TRC105) to CD105
Drug: Bevacizumab — Bevacizumab will be dosed every two weeks.
  Other Names: Avastin

SUMMARY:
The purpose of the study is to determine the overall response rate of single agent TRC105 and the combination of TRC105 and bevacizumab in patients with refractory GTN (including choriocarcinoma, placental site trophoblastic tumor (PSTT), and epithelioid trophoblastic tumor (ETT)). Up to 30 patients will be treated.

DETAILED DESCRIPTION:
TRC105 is a monoclonal antibody that binds to endoglin, an angiogenic target highly expressed on the tumor vessels and tumor cells in gestational trophoblastic neoplasia (GTN). Bevacizumab is a monoclonal antibody to vascular endothelial growth factor (VEGF) that inhibits angiogenesis and extends survival in patients with a wide variety of solid tumor types. TRC105 has been well tolerated as a single agent and when combined with bevacizumab. These antibodies may be efficacious in refractory GTN, a tumor type that is highly vascular and has been shown to densely express endoglin.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to consent for self to participate in study
2. Willingness and ability to comply with study procedures
3. Elevated serum hCG (in cases of choriocarcinoma); elevated hCG or measurable disease (in cases of PSTT or ETT)
4. Histologically proven trophoblastic neoplasia, or clinically demonstrated trophoblastic neoplasia that has progressed following treatment with at least one chemotherapy regimen that included 2 or more chemotherapy agents.
5. Age of 16 years or older
6. ECOG performance status ≤ 1
7. Resolution of all acute adverse events resulting from prior cancer therapies to NCI CTCAE grade ≤ 1 or baseline
8. Adequate organ function

Exclusion Criteria:

1. Male
2. Prior treatment with TRC105
3. . Current treatment on another therapeutic clinical trial
4. Uncontrolled chronic hypertension defined as systolic > 150 or diastolic > 90 despite optimal therapy
5. Significant pericardial effusion, pleural effusion, or ascites
6. Active bleeding or pathologic condition that carries a high risk of bleeding
7. Tumors located in the central chest or other location where bleeding is associated with high morbidity
8. Thrombolytic use (except to maintain i.v. catheters) within 10 days prior to first day of study therapy
9. Angina, MI, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) within the past 6 months. Deep venous thrombosis within 6 months, unless the patient is therapeutically anti-coagulated for at least 2 weeks. In this situation, low molecular weight heparin is preferred
10. Known active viral or nonviral hepatitis
11. Pregnant or actively breastfeeding without intention to discontinue prior to initiation of study
12. Open wounds or unhealed fractures within 28 days of starting study treatment
13. History of peptic ulcer disease or erosive gastritis within the past 6 months, unless treated for the condition and complete resolution has been documented by esophagogastroduodenoscopy (EGD) within 28 days of starting study treatment
14. History of gastrointestinal perforation or fistula in the past 6 months, or while previously on antiangiogenic therapy, unless underlying risk has been resolved
15. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
16. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study
17. History of brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease. Patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been administered for brain edema for at least 28 days
18. Receipt of systemic anticancer therapy, including investigational agents, within 28 days of starting study treatment. If anticancer therapy was given within 28 days of starting study treatment, patients may be included if 5 times the elimination half-life of the drug has passed
19. Patients who have received wide field radiotherapy ≤ 28 days (defined as > 50% of volume of pelvic bones or equivalent) or limited field radiation for palliation < 14 days prior to starting study treatment or those patients who have not recovered adequately from side effects of such therapy
20. Major surgical procedure or significant traumatic injury within 6 weeks prior to study registration or not fully recovered from any such procedure

Ages: 16 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Theuer, MD, PhD, Study Director — Tracon Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Ohio State University, Columbus, Ohio
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRC105 and/or Bevacizumab
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TRC105 and/or Bevacizumab
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 48 [46 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3
Number of Prior Regimens [Median (Full Range); unit: prior regimens] | 6 [1 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate on TRC105 Alone and on the Combination of TRC105 and Bevacizumab
Description: Antitumor Activity of Single Agent TRC105 and the Combination of TRC105 and Bevacizumab will be assessed via RECIST 1.1 and by measuring circulating bHCG. Disease progression is defined as >20% increase (the absolute increase must be ≥10 IU/L) above the nadir on consecutive measurements separated by at least two weeks; Partial response is defined as a hCG decrease of 50% or more from starting value on consecutive measurements; Complete response will be defined as normalization of hCG on consecutive measurements separated by at least two weeks; Stable disease will be defined as the absence of response or progression on 3 consecutive measurements separated by at least two weeks.
Time Frame: 8 weeks
Population: All patients who had a baseline scan and at least 1 on study assessment
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 and/or Bevacizumab
Number analyzed (Participants) | 3
Participants
  Number of patients with best response of PR | 0
  Number of patients with best response of SD | 0
  Number of patients with best response of PD | 3
  Number of patients with best response of CR | 0

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Median Progression-Free Survival (PFS) via Serum hCG levels and response evaluation according to RECIST version 1.1 as a preliminary measure of the antitumor activity of TRC105. Disease progression is defined as >20% increase (the absolute increase must be ≥10 IU/L) above the nadir on consecutive measurements separated by at least two weeks; Partial response is defined as a hCG decrease of 50% or more from starting value on consecutive measurements; Complete response will be defined as normalization of hCG on consecutive measurements separated by at least two weeks; Stable disease will be defined as the absence of response or progression on 3 consecutive measurements separated by at least two weeks. Patients must have screening (baseline) and at least one on study CT scan to be considered evaluable.
Time Frame: 8 weeks
Population: Progression Free Survival
Measure: Median (Full Range); unit: weeks
Arm/Group | TRC105 and/or Bevacizumab
Number analyzed (Participants) | 1
weeks | 6 [6 to 6]

3. Secondary Outcome: Overall Response Rate on Bevacizumab Alone
Description: Overall Response Rate on bevacizumab alone according to RECIST 1.1 in combination with serum hCG levels. Disease progression is defined as >20% increase (the absolute increase must be ≥10 IU/L) above the nadir on consecutive measurements separated by at least two weeks; Partial response is defined as a hCG decrease of 50% or more from starting value on consecutive measurements; Complete response will be defined as normalization of hCG on consecutive measurements separated by at least two weeks; Stable disease will be defined as the absence of response or progression on 3 consecutive measurements separated by at least two weeks.
Time Frame: 8 weeks
Population: No patients received bevacizumab alone.
Arm/Group | TRC105 and/or Bevacizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of TRC105.
Description: Mean serum TRC105 concentrations were assessed at cycle 1 and cycle 2 on day 1, 8, 15, and 22 and on day 1 of every subsequent cycle using validated methods in order to determine the Cmax of TRC105
Time Frame: cycle 2 day 1 (28 days after initiation of dosing)
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | TRC105 and/or Bevacizumab
Number analyzed (Participants) | 2
ng/mL | 232500 [199000 to 266000]

5. Secondary Outcome: TRC105 Immunogenicity as Assessed by Anti-Product Antibody (APA).
Description: Anti-Product Antibody (APA) concentrations will be measured using validated ELISA methods at the time points specified in the protocol. APA concentrations will be evaluated in the context of pharmacokinetic parameters and AE profiles. Number of patients with positive APA titers on study will be reported.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 and/or Bevacizumab
Number analyzed (Participants) | 3
Participants
  Number of patients with negative APA | 1
  Number of patients with positive APA | 2

6. Secondary Outcome: Frequency and Severity of Adverse Events
Description: Determine frequency and severity of adverse events as assessed by NCI CTCAE (Version 4.03)
Time Frame: 20 months
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 and/or Bevacizumab
Number analyzed (Participants) | 3
Participants
  Participants who experienced an SAE | 1
  Participants who experienced a TRC105 related SAE | 0

ADVERSE EVENTS:
Time Frame: Patients were followed for at least 28 days after the last dose of TRC105 study drug for adverse events, up to approximately 2 years.
Arm/Group | TRC105 and/or Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 and/or Bevacizumab (N=3)
Urinary Tract Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 and/or Bevacizumab (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 (7)
Ascites (Gastrointestinal disorders) | 1 (1)
Blood Amylase Increased (Investigations) | 1 (2)
Candiduria (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Faecal Incontinence (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 1 (2)
Fungal Test Positive (Investigations) | 1 (1)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Lipase Increased (Investigations) | 1 (2)
Localised Oedema (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Pelvic Abscess (Infections and infestations) | 1 (3)
Pyrexia (General disorders) | 1 (3)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (2)
Spinal Cord Compression (Nervous system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (2)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT02664961/SAP_000.pdf
  • Study Protocol (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT02664961/Prot_001.pdf